CLINICAL TRIAL: NCT04543747
Title: Mechanical Circulatory Support Korea Post Market Surveillance Study (MCS Korea PMS)
Brief Title: Mechanical Circulatory Support Korea Post Market Surveillance Study (PMS)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MCS Korea PMS
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: End-stage Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients implanted with HVAD System: Patients who require treatment with HVAD for use as bridge to cardiac transplantation (BTT) or destination therapy (DT) within the re-examination period are eligible for enrollment into the MCS Korea PMS. Patient consent may be obtained prior to HVAD implant or after receiving HVAD implant. Waiver of consent may be allowed if allowed by site's Institutional Review Board (IRB) or Ethics Committee (EC).
  Interventions: Device: HeartWare Ventricular Assist Device

INTERVENTIONS:
Device: HeartWare Ventricular Assist Device — The Medtronic HVAD® System is comprised of three major components: the HVAD Pump with inflow and outflow conduits, a Controller and power sources. In addition to these components, the system includes a Monitor, Battery Charger, AC and DC power adapters, and a Carrying Case. The HVAD® System is indicated for hemodynamic support in patients with advanced, refractory left ventricular heart failure; either as a bridge to cardiac transplantation (BTT), myocardial recovery, or as destination therapy (DT) in patients for whom subsequent transplantation is not planned.
  Other Names: HVAD

SUMMARY:
Medtronic is sponsoring this Mechanical Circulatory Support (MCS) Korea Post-Market Surveillance (PMS) to evaluate the safety and performance of the HeartWare Ventricular Assist Device System (HVAD® System) when used in routine clinical care practice in Korea. The MCS Korea PMS is conducted within Medtronic's Product Surveillance Platform (PSR).

DETAILED DESCRIPTION:
The MCS Korea PMS is an observational study conducted at two sites. This MCS Korea PMS is required by the Ministry of Food and Drug Safety (MFDS) as a condition of product approval according to Regulation on Medical Device Re-examination. The designated re-examination period is seven years after the approval date (06 Dec 2013 ~ 05 Dec 2020). All patients who require treatment of a commercially available HVAD System for approved indications between the designated re-examination period at a participating PSR site are eligible for enrollment. All enrolled patients will be followed until patient death, transplant, explant (where applicable), or the end of the study, on 05 Dec 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible product
* Patient is consented within the enrollment window or waiver of consent is approved

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results (i.e. no required intervention that could affect interpretation of all-around product safety and or effectiveness)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who require treatment with a HVAD for use as a bridge to cardiac transplantation (BTT) or a destination therapy (DT) within the re-examination period are eligible for enrollment into the MCS Korea PMS.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Survival rate up to 6 months and 24 months post-implant | Implant to 6 months, 24 months
  Success (or survival) will be defined as survival, heart transplantation, or explantation for recovery at 6 months post-implant for BTT patients, survival at 24 months post-implant for DT patients.

SECONDARY OUTCOMES:
Quality of life, as measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ), up to 24 months post-implant | Implant up through 24 months
  Characterize changes in quality of life over time
Functional status, as measured by the New York Heart Association (NYHA) classification, up to 24 months post-implant | Implant up through 24 months
  Characterize changes in NYHA class over time
Functional status, as measured by the 6-minute walk test, up to 24 months post-implant | Implant up through 24 months
  Characterize changes in 6-min walk test results (walked distance in meters) over time

OTHER OUTCOMES:
INTERMACS-defined Adverse Events up to 24 months post-implant | Implant to 24 months
  Summarize adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No